CLINICAL TRIAL: NCT03974035
Title: Does it Worth to Reinforce With Additional Anesthesia to Improve Postoperative Course After Orthognathic Surgery?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Servei Central d'Anestesiologia (Other)
Responsible Party: Principal Investigator, Gloria Molins Ballabriga, Principal Investigator, Servei Central d'Anestesiologia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1TDGM
Record Dates: First submitted 2019-05-13; First posted 2019-06-04 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Dentofacial Deformities
Keywords: Local anesthesia; Ropivacaine
MeSH Terms: conditions — Dentofacial Deformities | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: The investigators propose a double-blinded prospective comparative experimental study (patient and nurse). After the approval of the ethics committee of our hospital and the signed consent from each of the patients in the study, patients will be scheduled for bimaxillary osteotomy and will be randomly and prospectively assigned to one of the two groups with a plan to register up to 52 patients. Patients will not know the group that they have been assigned consecutively; and both the postoperative resuscitation nurses and the hospitalization nurses who will perform VAS records, opioid consumption, PONV and postoperative complications, will also be unaware of the analgesic treatment that the patient has received in the operating room. Patients will be assigned randomly to one group or another:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients undergoing elective bimaxillary osteotomy who receive a preincisional infiltration of lidocaine and adrenaline.
- Study Group (Experimental): Patients undergoing elective bimaxillary osteotomy who receive two infiltrations (firstly pre-incision with lidocaine and adrenaline, secondly pre-extubation with ropivacaine).
  Interventions: Drug: Second infiltration pre-extubation with ropivacaine

INTERVENTIONS:
Drug: Second infiltration pre-extubation with ropivacaine — The surgeon will proceed firstly with pre-incisional infiltration with lidocaine and adrenaline after intubation, and secondly with pre-extubation infiltration with ropivacaine at the intraoral and intranasal submucosal level in the maxilla and jaw to block the terminal branches of the maxillary and mandibular nerve
  Arms: Study Group

SUMMARY:
Bimaxillary osteotomy is a surgery procedure of the orthognathic surgery field for correction of dental and facial abnormalities, for both functional and aesthetic cases. The incidence of this abnormality is 5-10% of the population, and the etiology is unknown, with genetic, environmental and embryonic factors related. The surgery technic is complex, and requires osteotomy of the maxilla and jaw, which allows toward, forward, impact and rotation of these bones to fix the edges of the face. The anesthetic management of these patients is a challenge because of the difficult airway management and the perioperative pain control. Multimodal approach for pain control is a fact, and the use of local anesthesia is mandatory. The investigators propose the infiltration of local anesthesia in two different times, first pre-incision and second before awaking the patient, for a proper control of postoperative pain

DETAILED DESCRIPTION:
Bimaxillary osteotomy is a surgical procedure in the field of orthognathic surgery (from Latin, "ortho" straight and "gnatho" jaw) for the correction of dentofacial deformities, both for functional and aesthetic reasons. The incidence of this deformity is estimated to be around the 5-10% of the population. Genetic, environmental and embryonic factors are postulated to be the origin of such deformity, though its origin is still unknown. The surgical technique is complex, with the performance of mandibular and upper jaw osteotomies that allow to advance, retrude, impact and rotate these bones, to align the facial axes. For all these reasons, the anesthetic management of these patients is a challenge. First, the foreseeable difficulty of managing the patient's airway; and second, the control of the patient's pain in the perioperative period.

Therefore, bimaxillary osteotomy is a frequent surgery and potentially painful in adults. Bimaxillary surgery under general anesthesia is the common practice. And peripheral non-ultrasound-guided peripheral nerve blocks are widely used by surgeons. These minor blockades are used to avoid the undesired effects of anesthetics and analgesics; mainly the adverse respiratory effects of opioids. The practice of loco-regional anesthesia provides a control of perioperative pain in a multimodal way showing effective postoperative analgesia and minimizing the respiratory depression caused by the excess use of opioids.

In general, during bimaxillary surgery the surgeon performs the infiltrations with local anesthetic (LA) in a pre-incisional manner for the blockade of the terminal branches of the maxillary and mandibular nerve intranasally and intraorally. The choice of LA is influenced by considerations such as the start of action, duration and toxicity. A wide range of LA has been used in maxillofacial surgery, such as lidocaine and ropivacaine among others. Both LA produce a reversible blockade of the sodium channel of the neuronal membrane, and are synthetic derivatives of cocaine. Both possess three essential functional units (hydrophilic tertiary amide chain, linked by an intermediate amide chain, to another lipophilic aromatic ring-portion). This means, both LA are amide type; but even if they belong to the same group of LA there is still great differences in the beginning of action, duration of action and toxicity. Lidocaine has a faster start of action (short latency) than ropivacaine, and has an antiarrhythmic effect. Ropivacaine is more potent, the action last longer than lidocaine, has vasoconstrictor effect by itself and is less cardiotoxic than other equipotent LA such as bupivacaine and levobupivacaine.

The investigators avoid the use of a combination of LA for maxillary and mandibular nerve block. The combination of several local anesthetics in the same nerve block is sometimes used in perioperative anesthesia with the intention of compensating the short duration of action of some agents whose start of action is fast, such as lidocaine, and the high latency of the agents that present a more lasting action, such as ropivacaine. The combination of lidocaine and ropivacaine offers clinical advantages (rapid onset, long duration). However, to date, indications for combining LA are scarce because of the use of catheters in many forms of regional anesthesia that allow to prolong the duration of the block. This is nevertheless not an extended practice among anesthesiologists in maxillofacial surgery. On the other hand, it is important to also remember avoiding the use of maximum doses of two LA combined, which is based on the erroneous belief that their toxicities are independent; on the contrary, the toxicities have an additive character.

Multiple drugs have been used to increase the time of action of LA, such as adrenaline, clonidine, dexamethasone, ketamine and dexmedetomidine, among others. In the investigator's patients, adrenaline is always administered along with physiological serum pre-incision by the surgeon at the local level to improve the surgical field. The use of clonidine is ruled out because it is not supplied in the hospital center where the researchers will carry out the study. The use of dexamethasone and ketamine is ruled out, because they will be administered intravenously in the patient's perioperative period as anti-inflammatory agents and anesthetic adjuvant, respectively. And the use of dexmedetomidine is also ruled out in order to prolong the effect of the nerve blockade as this indication is not in the technical file.

Thus, the investigators propose to use firstly lidocaine and adrenaline pre-incision (antiarrhythmic effect and short duration of action). And secondly, they propose to use ropivacaine without adjuvant before extubation (vasoconstrictor effect and longer duration of action).

The control of postoperative pain is a primary factor to achieve greater patient satisfaction, better rehabilitation and shorter hospital stay. The current clinical guidelines recommend the management of postoperative pain control in a multimodal manner; and this includes the use of local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo scheduled bimaxillary surgery

Exclusion Criteria:

* patients who are scheduled for bimaxillary surgery together with another complementary surgical procedure (such as mentoplasty, rhinoplasty, blepharoplasty)
* age <18 years
* reinterventions
* urgent surgeries
* allergies to local anesthetics
* allergies to anti-inflammatories agents
* allergies to opioids
* American Society of Anesthesiology Physical Status Examination System (ASA) >3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Pain assessed by the visual analogue scale (VAS) in the immediate postoperative period | 2 hours postoperatively
  The main objective of the study is the evaluation of the effect of a peripheral pre-incisional minor nerve block with the use of a single local anesthetic (lidocaine), compared with the same nerve block in two times with different local anesthetics (lidocaine-preincisional and ropivacaine-pre-extubation), on the postoperative pain of patients undergoing elective bimaxillary osteotomy, evaluated by means of the visual analogue scale (VAS) of pain in the immediate postoperative period (2 hours postoperatively).
  The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patient is asked to mark their current pain level on the line. The examiner scores the VAS by measuring the distance in centimeters (0 to 10) from the "no pain" anchor point.

SECONDARY OUTCOMES:
Pain assessed by VAS at 4, 8 and up to 18 hours after surgery. | 4, 8 and up to 18 hours after surgery
  The comparison of visual analogue scale (VAS) of pain at 4, 8 and up to 18 hours after surgery.
  The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patient is asked to mark their current pain level on the line. The examiner scores the VAS by measuring the distance in centimeters (0 to 10) from the "no pain" anchor point.
Opioid use of rescue (intravenous methadone milligrams) | 2 and 18 hours postoperatively
  The comparison of the opioid use of rescue (intravenous methadone milligrams) in the immediate postoperative period in resuscitation (2 hours postoperatively) and in the hospitalization floor (18 hours postoperatively)
Postoperative nausea and vomiting (PONV) | 2 and 18 hours postoperatively
  Comparing the incidence of postoperative nausea and vomiting (PONV) in the immediate postoperative period in resuscitation and up to 18 hours after the surgery in the two groups of patients
Complications derived from the two infiltrations | Through surgery completion and 0 to 18 hours postoperatively
  Registry of complications derived from the two infiltrations

CONTACTS AND LOCATIONS:
Overall Officials: Federico Hernández-Alfaro, MD, DDS, PhD, Study Director — Instituto Maxilofacial - Centro Médico Teknon; Miriam DeNadal, MD, PhD, Study Director — Hospital Valle de Hebrón
Locations (1):
- Centro Medico Teknon - Grupo Quirón Salud, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of the study completion
Access Criteria: data access requests will be reviewed by an external independent Review Panel. Requestors will be required to sign a Data Access Agreement

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT03974035/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT03974035/ICF_001.pdf